CLINICAL TRIAL: NCT03108924
Title: An Open-Label, Single-Dose Study to Investigate the Influence of Renal Insufficiency on the Pharmacokinetics of MK-7264
Brief Title: The Pharmacokinetics of Gefapixant (MK-7264) in Participants With Renal Insufficiency (MK-7264-026)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7264-026; MK-7264-026-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Results first posted 2019-08-02 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Gefapixant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Moderate RI (Experimental): Participants with moderate renal insufficiency (RI) are treated with a single 50 mg dose of gefapixant
  Interventions: Drug: Gefapixant
- Severe RI (Experimental): Participants with severe RI are treated with a single 50 mg dose of gefapixant
  Interventions: Drug: Gefapixant
- Healthy Matched Controls (Other): Healthy, participants matched for age and body weight are treated with a single 50 mg dose of gefapixant
  Interventions: Drug: Gefapixant
- ESRD Requiring HD (Experimental): Participants with end stage renal disease (ESRD) requiring hemodialysis (HD), are treated in Period 1 with a single 50 mg dose of gefapixant immediately after the scheduled HD, followed in Period 2 with a single 50 mg dose of gefapixant two hours prior to HD. Between the Periods 1 and 2 MK-7264 dose administrations there was approximately a 7-day washout period with 3 dialysis sessions.
  Interventions: Drug: Gefapixant

INTERVENTIONS:
Drug: Gefapixant — After an overnight fast participants receive a single oral dose of 50 mg gefapixant, in one 50 mg tablet.
  Other Names: MK-7264

SUMMARY:
This trial aims to evaluate the plasma pharmacokinetics of gefapixant (MK-7264) administered to participants with varying degrees of renal insufficiency (RI) compared to healthy matched controls; and to investigate the extent of MK-7264 removal by hemodialysis (HD) in participants with end stage renal disease (ESRD), following administration of a single 50 mg dose of gefapixant.

ELIGIBILITY:
Inclusion Criteria:

* Is a non-smoker or moderate smoker (≤ 20 cigarettes/day or the equivalent) who agrees to consume no more than 10 cigarettes or equivalent/day from the time of screening and throughout the period of sample collection.
* Has a body mass index (BMI) ≥ 18.5 and ≤ 40.0 kg/m^2,
* Is judged to be in good health based on medical history, physical examination, vital signs, and laboratory safety tests. Has no clinically significant electrocardiogram (ECG) abnormality, as deemed by the Investigator.
* Females are non-pregnant, and non-breast feeding. If female with reproductive potential, they must demonstrate they are not pregnant and agree to use (and/or have their partner use) two (2) acceptable methods of birth control beginning at screening, throughout the study and until 2 weeks after dosing of study drug.
* Participants with ESRD requiring HD has been maintained on stable regimen of thrice-weekly HD for at least 3 months prior to first dosing.
* Healthy participants, must be within ± 10 years of the mean age of participants with RI; and must be within ± 10 kg of the mean weight of participants with RI.

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit, or expected during the conduct of the study.
* Has a history or presence of clinically significant medical or psychiatric condition or disease.
* Has a history of any illness that, in the opinion of the Investigator, might confound the results of the study or poses an additional risk by participating in the study.
* Has a history or presence of alcoholism or drug abuse within the past 6 months prior to dosing.
* Has a history or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds (including sulfonamides).
* Has a history or presence of renal artery stenosis; or major risk factors for renal/urinary calculi.
* Has rapidly fluctuating renal function as determined by historical measurements.
* Female who is pregnant, or lactating.
* Has positive results for urine or saliva drug and/or urine or breath alcohol at screening or check-in.
* Is positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Has positive macroscopic hematuria or crystalluria at screening or check-in.
* Is unable to refrain from or anticipates using any medication or substance including prescription or over-the-counter, vitamin supplements, natural or herbal supplements.
* Has been on a diet incompatible with the on-study diet, within the 28 days prior to dosing.
* Has donated blood or had significant blood loss within 56 days prior to dosing.
* Has donated plasma within 7 days prior to dosing.
* Has taken gefapixant at any time prior to dosing on the current study.
* Has participated in another clinical trial within 28 days prior to dosing based on the latest blood collection or dosing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-09-03 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami ( Site 0001), Hialeah, Florida
  - Orlando Clinical Research Center ( Site 0002), Orlando, Florida

REFERENCES:
- [Result] Nussbaum JC, Hussain A, Min KC, Marbury TC, Lasseter K, Stoch SA, Iwamoto M. Effects of Renal Impairment on the Pharmacokinetics of Gefapixant, a P2X3 Receptor Antagonist. J Clin Pharmacol. 2022 Nov;62(11):1435-1444. doi: 10.1002/jcph.2094. Epub 2022 Jul 7. PMID 35656754

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, 2-part, single dose study. In Part 1, MK-7264 was evaluated in participants with moderate and severe renal impairment (RI) compared to healthy matched control participants. In Part 2, MK-7264 was evaluated in 2 periods in participants with end stage renal disease (ESRD) requiring hemodialysis (HD).
Groups:
- [Part 1] Moderate RI: Participants with moderate renal impairment (RI) received a single oral dose of gefapixant 50 mg
- [Part 1] Severe RI: Participants with severe RI received a single oral dose of gefapixant 50 mg
- [Part 2] ESRD: Participants with ESRD requiring HD received a single oral dose of gefapixant 50 mg immediately after HD in Period 1, followed by a single oral dose of gefapixant 50 mg two hours prior to HD in Period 2. Between the Periods 1 and 2 MK-7264 dose administrations there was approximately a 7-day washout period with 3 dialysis sessions.
- [Part 1 and Part 2] Healthy Controls: Healthy participants were matched to participants with moderate and severe RI (Part 1) and participants with ESRD (Part 2).
Period: Overall Study
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2] ESRD | [Part 1 and Part 2] Healthy Controls
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- [Part 1] Moderate RI: Participants with moderate RI received a single oral dose of gefapixant 50 mg
- Total: Total of all reporting groups
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2] ESRD | [Part 1 and Part 2] Healthy Controls | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (10.76) | 64.3 (5.75) | 52.7 (7.12) | 65.8 (5.00) | 62.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 1 | 4
  Male | 5 | 4 | 6 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 2 | 12
  Not Hispanic or Latino | 2 | 2 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 4 | 3 | 9
  White | 4 | 6 | 2 | 3 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: [Parts 1 and 2] Mean Area Under the Concentration-Time Curve From Time Zero Up to Infinity (AUC0-inf) of Gefapixant 50 mg (Categorical Analysis)
Description: The mean area under the concentration-time curve from time 0 to infinity (AUC0-inf) of plasma gefapixant was assessed. In Part 1, participants with Moderate RI, Severe RI, or normal renal function (i. e., Healthy Controls) received a single oral dose of gefapixant 50 mg at Hour 0 on Day 1. In Part 2, Period 1, ESRD participants received a single oral dose of gefapixant 50 mg at Hour 0 on Day 1, immediately following the scheduled HD. In Part 2, Period 2, participants received a single oral dose of gefapixant 50 mg at Hour 0 on Day 1, approximately 2 hours prior to initiation of HD. Non-model based summary statistics were provided for the number of participants with non-missing data, as well as mean and standard deviation values. Serial blood samples for the determination of plasma gefapixant concentrations were collected at predose and at selected time points over 72 hours postdose.
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. The ESRD Non-HD and ESRD HD arms are a split of the original ESRD arm. The same 6 participants are in both Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- [Part 2, Period 1] ESRD Non-HD: Participants with ESRD requiring HD, but not on HD, received a single oral dose of gefapixant 50 mg immediately after the scheduled HD, in Period 1
- [Part 2, Period 2] ESRD HD: Participants with ESRD requiring HD, and on HD, received a single oral dose of gefapixant 50 mg two hours prior to HD in Period 2. Between gefapixant dose administrations in Periods 1 and 2, there was approximately a 7-day washout period with 3 dialysis sessions.
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD | [Part 1 and Part 2] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 6450 (1910) | 9970 (4080) | 9990 (3610) | 8590 (4190) | 2280 (1160)

2. Primary Outcome: [Part 2] Geometric Least Squares Mean (GM) AUC0-inf in ESRD HD Participants vs. ESRD Non-HD Participants (Categorical Analysis)
Description: To evaluate the extent of gefapixant removal by hemodialysis, individual values of AUC0-inf, were natural log (ln)-transformed and analyzed using a linear mixed-effects model with population (ESRD Non-HD, ESRD HD) as a fixed effect. An unstructured covariance matrix was used to allow for unequal variances and to model the correlation between the 2 measurements within each participant. A two-sided 90% confidence interval (CI) for the true difference in means was calculated for AUC0-inf. These confidence limits were exponentiated to obtain the 90% CI for the geometric least squares mean ratio (GMR) (ESRD HD/ESRD Non-HD) for AUC0-inf.
Time Frame: Part 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 2 who were compliant with the study procedure and had available data were included. A single participant with 6 missing plasma samples in Part 2, Period 1 was excluded from the ESRD Non-HD group. The ESRD Non-HD and ESRD HD arms are a split of the original ESRD arm. The same 6 participants were in Periods 1 and 2.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD
Number analyzed (Participants) | 5 | 6
ng*hr/mL | 10100 [6300 to 16200] | 7810 [4740 to 12900]
Statistical Analysis 1: Comparison: [Part 2, Period 1] ESRD Non-HD vs [Part 2, Period 2] ESRD HD; Test type: Other; Categorical Analysis; GMR = 0.77, 90% CI 2-sided [0.53 to 1.13] — GMR = GM for ESRD HD / GM for ESRD Non-HD

3. Primary Outcome: [Part 1] Estimated AUC0-inf of Gefapixant 50 mg in Participants With Body Surface Area (BSA)-Normalized Estimated Glomerular Filtration Rate (eGFR) (Regression Analysis)
Description: AUC0-inf values of plasma gefapixant based on BSA-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of AUC0-inf were natural log-transformed and evaluated with a linear fixed-effects model containing BSA-normalized eGFR as a continuous variable. The back transformed mean AUC0-inf and corresponding 95% CI were predicted at the midpoint of the BSA enormalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 1 who were compliant with the study procedure and had available data were included.
Measure: Mean (95% Confidence Interval); unit: ng*hr/mL
Groups:
- [Part 1] Healthy Controls: Healthy participants were matched to participants with moderate and severe RI (Part 1).
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 6350 [5210 to 7750] | 8580 [6710 to 11000] | 2280 [1700 to 3050]

4. Primary Outcome: [Part 1] Estimated AUC0-inf of Gefapixant 50 mg in Participants With BSA Non-Normalized eGFR (Regression Analysis)
Description: AUC0-inf values of plasma gefapixant based on BSA non-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of AUC0-inf were natural log-transformed and evaluated with a linear fixed-effects model containing BSA non-normalized eGFR as a continuous variable. The back transformed mean AUC0-inf and corresponding 95% CI were predicted at the midpoint of the BSA non-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their BSA non-normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 1 who were compliant with the study procedure and had available data were included. For non-normalized eGFR estimates, participants originally assigned to the severe RI group were reassigned: 1 participant reassigned to the mild RI group (excluded from analysis), and 1 participant reassigned to the moderate RI group.
Measure: Mean (95% Confidence Interval); unit: ng*hr/mL
Groups:
- [Part 1] Healthy Controls: Healthy Control participants received a single oral dose of gefapixant 50 mg
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 7 | 4 | 6
ng*hr/mL | 6850 [5580 to 8410] | 8840 [6900 to 11300] | 2370 [1790 to 3130]

5. Primary Outcome: [Part 1 and 2] Estimated AUC0-inf of Gefapixant 50 mg in Participants With Moderate RI, Severe RI, ESRD Non-HD, or Normal Renal Function (Categorical Analysis)
Description: Geometric mean and 95%CI for AUC0-inf were estimated in participants with moderate RI, severe RI, ESRD requiring but not receiving HD, and normal renal function (i. e., Healthy Controls). Individual values of AUC0-inf, were ln-transformed and evaluated with a linear fixed-effects heterogeneous variance model containing a categorical effect for population (ESRD Non-HD, severe RI, moderate RI, and healthy matched control, based on BSA normalized eGFR). To compare subjects with RI in each of the renal categories to subjects with normal renal function, a two-sided 90% CI for the true difference in means (renal impairment - normal renal function) was calculated for AUC0-inf, using the mean square error from the model and referencing a t-distribution. For each of the RI populations, these confidence limits were exponentiated to obtain the 90% CI for the GMR (renal impairment/normal renal function).
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 were compliant with the study procedure and had available data were included. A single participant with 6 missing plasma samples in Part 2, Period 1 was excluded from the ESRD Non-HD group. The same 6 participants were in Periods 1 and 2.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 5 | 6
ng*hr/mL | 6230 [4610 to 8400] | 9270 [5940 to 14500] | 9900 [5940 to 16500] | 2090 [1320 to 3310]
Statistical Analysis 1: Comparison: [Part 1] Moderate RI; Test type: Other; Categorical Analysis; GMR = 2.98, 90% CI 2-sided [2.01 to 4.41] — GMR = GM for Moderate RI / GM for Healthy Controls
Statistical Analysis 2: Comparison: [Part 1] Severe RI; Test type: Other; Categorical Analysis; GMR = 4.43, 95% CI 2-sided [2.82 to 6.96] — GMR = GM for Severe RI / GM for Healthy Controls
Statistical Analysis 3: Comparison: [Part 2, Period 1] ESRD Non-HD; Test type: Other; Categorical Analysis; GMR = 4.74, 90% CI 2-sided [2.95 to 7.59] — GMR = GM for ESRD HD / GM for Healthy Controls

6. Primary Outcome: [Parts 1 and 2] Mean Area Under the Concentration-Time Curve of From Time Zero to the Last Quantifiable Sample (AUC0-last) of Gefapixant 50 mg
Description: The mean area under the concentration-time curve from time 0 to the last quantifiable sample (AUC0-last), above the lower limit of quantitation (LLOQ), of plasma gefapixant in participants with moderate RI, severe RI, ESRD, or normal renal function (i. e., Healthy Controls) was assessed. Non-model based summary statistics were provided for the number of participants with non-missing data, as well as mean and standard deviation values.
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 5930 (1950) | 7630 (3080) | 7790 (2740) | 6460 (2640) | 2000 (1230)

7. Primary Outcome: [Part 2] Geometric Least Squares Mean AUC0-last of Gefapixant 50 mg in ESRD HD Participants vs. ESRD Non-HD Participants (Categorical Analysis)
Description: To evaluate the extent of gefapixant removal by hemodialysis, individual values of AUC0-last, were ln-transformed and analyzed using a linear mixed-effects model with population (ESRD Non-HD, ESRD HD) as a fixed effect. An unstructured covariance matrix was used to allow for unequal variances and to model the correlation between the 2 measurements within each participant. A two-sided 90% CI for the true difference in means was calculated for AUC0-last. These confidence limits were exponentiated to obtain the 90% CI for the geometric least squares mean ratio (GMR) (ESRD HD/ESRD Non-HD) for AUC0-last.
Time Frame: Part 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 2 who complied with the study procedure and had available data were included. A single participant with 6 missing plasma samples in Part 2, Period 1 was excluded from the ESRD Non-HD group. The ESRD Non-HD and ESRD HD arms were split from the original ESRD arm. The same 6 participants were in Periods 1 and 2.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD
Number analyzed (Participants) | 5 | 6
ng*hr/mL | 7870 [5080 to 12200] | 6030 [3930 to 9260]
Statistical Analysis 1: Comparison: [Part 2, Period 1] ESRD Non-HD vs [Part 2, Period 2] ESRD HD; Test type: Other; Categorical Analysis; GMR = 0.77, 90% CI 2-sided [0.54 to 1.08] — GMR = GM for ESRD HD / GM for ESRD Non-HD

8. Primary Outcome: [Part 1] Estimated AUC0-last of Gefapixant 50 mg in Participants With BSA-Normalized eGFR (Regression Analysis)
Description: AUC0-last values of plasma gefapixant based on BSA-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of AUC0last were natural log-transformed and evaluated with a linear fixed-effects model containing BSA-normalized eGFR as a continuous variable. The mean AUC0-ilast and corresponding 95% CI were back-transformed and predicted at the midpoint of th BSA enormalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 1 who were compliant with the study procedure and had available data were included.
Measure: Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL | 5310 [4280 to 6590] | 7130 [5470 to 9300] | 1940 [1410 to 2660]

9. Primary Outcome: [Part 1] Estimated AUC0-last of Gefapixant 50 mg in Participants With BSA Non-Normalized eGFR (Regression Analysis)
Description: AUC0-last values of plasma gefapixant based on BSA non-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of AUC0-last were natural log-transformed and evaluated with a linear fixed-effects model containing BSA non-normalized eGFR as a continuous variable. The back transformed mean AUC0-last and corresponding 95% CI were predicted at the midpoint of the BSA non-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their BSA non-normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 7 | 4 | 6
ng*hr/mL | 5740 [4620 to 7120] | 7380 [5690 to 9580] | 2000 [1490 to 2680]

10. Primary Outcome: [Parts 1 and 2] Estimated AUC0-last of Gefapixant 50 mg in Participants With Moderate RI, Severe RI, ESRD Non-HD, or Normal Renal Function (Categorical Analysis)
Description: Geometric mean and 95%CI for AUC0-last were estimated in participants with moderate RI, severe RI, ESRD requiring but not receiving HD, and normal renal function (i. e., Healthy Controls). Individual values of AUC0-last, were ln-transformed and evaluated with a linear fixed-effects heterogeneous variance model containing a categorical effect for population (ESRD Non-HD, severe RI, moderate RI, and healthy matched control, based on BSA normalized eGFR). To compare subjects with RI in each of the renal categories to subjects with normal renal function, a two-sided 90% CI for the true difference in means (renal impairment - normal renal function) was calculated for AUC0-last, using the mean square error from the model and referencing a t-distribution. For each of the RI populations, these confidence limits were exponentiated to obtain the 90% CI for the GMR (renal impairment/normal renal function).
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. A single participant was excluded from the ESRD Non-HD group since this participant had 6 missing peripheral plasma samples in Part 2, Period 1.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 5 | 6
ng*hr/mL | 5670 [4050 to 7940] | 7170 [4800 to 10700] | 7770 [4840 to 12500] | 1760 [995 to 3100]
Statistical Analysis 1: Comparison: [Part 1] Moderate RI; Test type: Other; Categorical Analysis; GMR = 3.23, 90% CI 2-sided [2.01 to 5.20] — GMR = GM for Moderate RI / GM for Healthy Controls
Statistical Analysis 2: Comparison: [Part 1] Severe RI; Test type: Other; Categorical Analysis; GMR = 4.08, 90% CI 2-sided [2.49 to 6.70] — GMR = GM for Severe RI / GM for Healthy Controls
Statistical Analysis 3: Comparison: [Part 2, Period 1] ESRD Non-HD; Test type: Other; Categorical Analysis; GMR = 4.43, 90% CI 2-sided [2.65 to 7.39] — GMR = GM for ESRD Non-HD / GM for Healthy Controls

11. Primary Outcome: [Parts 1 and 2] Maximum Concentration (Cmax) of Gefapixant 50 mg
Description: The maximum concentration (Cmax) of plasma gefapixant in participants with moderate RI, severe RI, ESRD Non-HD, ESRD HD, or normal renal function (i. e., Healthy Controls) following administration of gefapixant 50 mg was assessed. Non-model based summary statistics were provided for the number of participants with non-missing data, as well as mean and standard deviation values. Serial blood samples for the determination of plasma gefapixant concentrations were collected at predose and at selected time points over 72 hours postdose.
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included in the primary analysis dataset at the end of the study. The ESRD Non-HD and ESRD HD arms are a split of the original ESRD arm. The same 6 participants were in both Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 338 (127) | 311 (137) | 281 (92.5) | 228 (87.1) | 173 (95.7)

12. Primary Outcome: [Part 2] Geometric Least Squares Mean Cmax of Gefapixant 50 mg in ESRD HD Participants vs. ESRD Non-HD Participants (Categorical Analysis)
Description: To evaluate the extent of gefapixant removal by hemodialysis, individual values of Cmax, were ln transformed and analyzed using a linear mixed-effects model with population (ESRD Non-HD, ESRD HD) as a fixed effect. An unstructured covariance matrix was used to allow for unequal variances and to model the correlation between the 2 measurements within each participant. A two-sided 90% CI for the true difference in means was calculated for Cmax. These confidence limits were exponentiated to obtain the 90% CI for the geometric least squares mean ratio (GMR) (ESRD HD/ESRD Non-HD) for Cmax.
Time Frame: Part 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 7
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD
Number analyzed (Participants) | 5 | 6
ng/mL | 292 [194 to 439] | 214 [142 to 322]
Statistical Analysis 1: Comparison: [Part 2, Period 1] ESRD Non-HD vs [Part 2, Period 2] ESRD HD; Test type: Other; Categorical Analysis; GMR = 0.73, 90% CI 2-sided [0.52 to 1.03] — GMR = GM for ESRD HD / GM for ESRD Non-HD

13. Primary Outcome: [Part 1] Estimated Cmax of Gefapixant 50 mg in Participants With BSA-Normalized eGFR (Regression Analysis)
Description: Cmax values of plasma gefapixant based on BSA-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of Cmax were natural log-transformed and evaluated with a linear fixed-effects model containing BSA-normalized eGFR as a continuous variable. The back transformed mean Cmax and corresponding 95% CI were predicted at the midpoint of the BSA enormalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their normalized eGFR estimates were predicted at midpoint 75 mL/min. Serial blood samples for the determination of plasma gefapixant concentrations were collected at predose and at selected time points over 72 hours postdose.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 1 who were compliant with the study procedure and had available data were included.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 272 [211 to 351] | 318 [233 to 435] | 160 [110 to 232]

14. Primary Outcome: [Part 1] Estimated Cmax of Gefapixant 50 mg in Participants With BSA Non-Normalized eGFR (Regression Analysis)
Description: Cmax values of plasma gefapixant based on BSA non-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of Cmax were natural log-transformed and evaluated with a linear fixed-effects model containing BSA non-normalized eGFR as a continuous variable. The back transformed mean Cmax and corresponding 95% CI were predicted at the midpoint of the BSA non-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their BSA non-normalized eGFR estimates were predicted at midpoint 75 mL/min. Serial blood samples for the determination of plasma gefapixant concentrations were collected at predose and at selected time points over 72 hours postdose.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 7 | 4 | 6
ng/mL | 286 [222 to 369] | 329 [242 to 447] | 160 [113 to 226]

15. Primary Outcome: [Part 1 and 2] Estimated Cmax of Gefapixant 50 mg in Participants With Moderate RI, Severe RI, ESRD Non-HD, or Normal Renal Function (Categorical Analysis)
Description: Geometric mean and 95%CI for Cmax were estimated in participants with moderate RI, severe RI, ESRD requiring but not receiving HD, and normal renal function (i. e., Healthy Controls). Individual values of Cmax, were ln-transformed and evaluated with a linear fixed-effects heterogeneous variance model containing a categorical effect for population (ESRD Non-HD, severe RI, moderate RI, and healthy matched control, based on BSA normalized eGFR). To compare subjects with RI in each of the renal categories to subjects with normal renal function, a two-sided 90% CI for the true difference in means (renal impairment - normal renal function) was calculated for Cmax, using the mean square error from the model and referencing a t-distribution. For each of the RI populations, these confidence limits were exponentiated to obtain the 90% CI for the GMR (renal impairment/normal renal function).
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All Parts 1 and 2 participants who were compliant with the study procedure and had available data were included. A single participant was excluded from the ESRD Non-HD group since this participant had 6 missing peripheral plasma samples in Part 2, Period 1.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 5 | 6
ng/mL | 316 [201 to 496] | 286 [178 to 458] | 287 [187 to 441] | 151 [82.8 to 277]
Statistical Analysis 1: Comparison: [Part 1] Moderate RI; Test type: Other; Categorical Analysis; GMR = 2.09, 90% CI 2-sided [1.22 to 3.56] — GMR = GM for Moderate RI / GM for Healthy Controls
Statistical Analysis 2: Comparison: [Part 1] Severe RI; Test type: Other; Categorical Analysis; GMR = 1.89, 95% CI 2-sided [1.10 to 3.25] — GMR = GM for Severe RI / GM for Healthy Controls
Statistical Analysis 3: Comparison: [Part 2, Period 1] ESRD Non-HD; Test type: Other; Categorical Analysis; GMR = 1.90, 90% CI 2-sided [1.13 to 3.19] — GMR = GM for ESRD Non-HD / GM for Healthy Controls

16. Primary Outcome: [Parts 1 and 2] Apparent Clearance (CL/F) of Gefapixant 50 mg
Description: The apparent clearance (CL/F) of plasma gefapixant after oral administration of gefapixant 50 mg in participants with moderate RI, severe RI, ESRD requiring HD, or normal renal function (i. e., Healthy Controls) was assessed. Non-model based summary statistics were provided for the number of participants with non-missing data, as well as mean and standard deviation values. Serial blood samples for the determination of plasma gefapixant concentrations were collected at predose and at selected time points over 72 hours postdose.
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. The ESRD Non-HD and ESRD HD arms were split from the original ESRD arm. The same 6 participants were in Periods 1 and 2.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L/hr | 8.30 (2.25) | 5.81 (2.47) | 5.67 (2.28) | 7.00 (3.09) | 25.7 (9.42)

17. Primary Outcome: [Part 2] Geometric Least Squares Mean CL/F of Gefapixant 50 mg in ESRD HD Participants vs. ESRD Non-HD Participants (Categorical Analysis)
Description: To evaluate the extent of gefapixant removal by hemodialysis, individual values of CL/F, were ln-transformed and analyzed using a linear mixed-effects model with population (ESRD Non-HD, ESRD HD) as a fixed effect. An unstructured covariance matrix was used to allow for unequal variances and to model the correlation between the 2 measurements within each participant. A two-sided 90% CI for the true difference in means was calculated for CL/F. These confidence limits were exponentiated to obtain the 90% CI for the geometric least squares mean ratio (GMR) (ESRD HD/ESRD Non-HD) for CL/F.
Time Frame: Part 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 2, Period 1] ESRD Non-HD | [Part 2, Period 2] ESRD HD
Number analyzed (Participants) | 5 | 6
L/hr | 4.95 [3.08 to 7.94] | 6.40 [3.89 to 10.6]
Statistical Analysis 1: Comparison: [Part 2, Period 1] ESRD Non-HD vs [Part 2, Period 2] ESRD HD; Test type: Other; Categorical Analysis; GMR = 1.30, 90% CI 2-sided [0.88 to 1.90] — GMR = GM for ESRD / GM for ESRD Non-HD

18. Primary Outcome: [Part 1] Estimated CL/F of Gefapixant 50 mg in Participants With BSA-Normalized eGFR (Regression Analysis)
Description: CL/F values of plasma gefapixant based on BSA-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of CL/F were natural log-transformed and evaluated with a linear fixed-effects model containing BSA-normalized eGFR as a continuous variable. The back transformed mean CL/F and corresponding 95% CI were predicted at the midpoint of the BSA enormalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Part 1 who were compliant with the study procedure and had available data were included.
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
L/hr | 7.87 [6.45 to 9.60] | 5.83 [4.56 to 7.45] | 21.9 [16.4 to 29.4]

19. Primary Outcome: [Part 1] Estimated CL/F of Gefapixant 50 mg in Participants With BSA Non-Normalized eGFR (Regression Analysis)
Description: CL/F values of plasma gefapixant based on BSA non-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of CL/F were natural log-transformed and evaluated with a linear fixed-effects model containing BSA non-normalized eGFR as a continuous variable. The back transformed mean CL/F and corresponding 95% CI were predicted at the midpoint of the BSA non-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their BSA non-normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Part 1 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 7 | 4 | 6
L/hr | 7.30 [5.95 to 8.96] | 5.66 [4.42 to 7.24] | 21.1 [16.0 to 27.9]

20. Primary Outcome: [Parts 1 and 2] Estimated CL/F of Gefapixant 50 mg in Participants With Moderate RI, Severe RI, ESRD Non-HD, or Normal Renal Function (Categorical Analysis)
Description: Geometric mean and 95% CI for CL/F were estimated in participants with moderate RI, severe RI, ESRD requiring but not receiving HD, and normal renal function (i. e., Healthy Controls). Individual values of CL/F, were ln-transformed and evaluated with a linear fixed-effects heterogeneous variance model containing a categorical effect for population (ESRD Non-HD, severe RI, moderate RI, and healthy matched control, based on BSA normalized eGFR). To compare subjects with RI in each of the renal categories to subjects with normal renal function, a two-sided 90% CI for the true difference in means (renal impairment - normal renal function) was calculated for CL/F, using the mean square error from the model and referencing a t-distribution. For each of the RI populations, these confidence limits were exponentiated to obtain the 90% CI for the GMR (renal impairment/normal renal function).
Time Frame: Parts 1 and 2 - Predose, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. A single participant with 6 missing plasma samples in Part 2, Period 1 was excluded from the ESRD Non-HD group.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2, Period 1] ESRD Non-HD | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 5 | 6
L/hr | 8.03 [5.95 to 10.8] | 5.40 [3.46 to 8.41] | 5.05 [3.03 to 8.42] | 23.9 [15.1 to 37.9]
Statistical Analysis 1: Comparison: [Part 1] Moderate RI; Test type: Other; Categorical Analysis; GMR = 0.34, 95% CI 2-sided [0.23 to 0.50] — GMR = GM for Moderate RI / GM for Healthy Controls
Statistical Analysis 2: Comparison: [Part 1] Severe RI; Test type: Other; Categorical Analysis; GMR = 0.23, 95% CI 2-sided [0.14 to 0.35] — GMR = GM for Severe RI / GM for Healthy Controls
Statistical Analysis 3: Comparison: [Part 2, Period 1] ESRD Non-HD; Test type: Other; Categorical Analysis; GMR = 0.21, 95% CI 2-sided [0.13 to 0.34] — GMR = GM for ESRD Non-HD / GM for Healthy Controls

21. Primary Outcome: [Parts 1 and 2] Renal Clearance (CLr) of Gefapixant 50 mg
Description: The renal clearance (CLr) in participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) was assessed. Non-model base summary statistics were provided. Renal clearance could not be assessed for participants with ESRD. Urine specimens were obtained by spot collection predose and at multiple timepoints postdose.
Time Frame: Parts 1 and 2 - Predose and at 0-12 hrs, 12-24 hrs, and 24-48 hrs post dose
Population: All participants who were compliant with the study procedure and had available data were included. Renal clearance could not be assessed for participants with ESRD.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
L/hr | 2.10 (0.522) | 0.755 (0.387) | 6.72 (1.28)

22. Primary Outcome: [Parts 1 and 2] Estimated CLr of Gefapixant 50 mg in Participants With Moderate RI, Severe RI, or Normal Renal Function (Categorical Analysis)
Description: Geometric mean and 95% CI for CLr were estimated in participants with moderate RI, severe RI, and normal renal function (i. e., Healthy Controls). Individual values of CLr, were ln-transformed and evaluated with a linear fixed-effects heterogeneous variance model containing a categorical effect for population (severe RI, moderate RI, and healthy matched control, based on BSA normalized eGFR). To compare subjects with RI in each of the renal categories to subjects with normal renal function, a two-sided 90% CI for the true difference in means (renal impairment - normal renal function) was calculated for CLr, using the mean square error from the model and referencing a t-distribution. For each of the RI populations, these confidence limits were exponentiated to obtain the 90% CI for the GMR (renal impairment/normal renal function).
Time Frame: Parts 1 and 2 - Predose and at 0-12 hrs, 12-24 hrs, and 24-48 hrs post dose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. Renal clearance could not be assessed for participants with ESRD.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
L/hr | 2.05 [1.59 to 2.65] | 0.680 [0.403 to 1.15] | 6.61 [5.34 to 8.17]
Statistical Analysis 1: Comparison: [Part 1] Moderate RI; Test type: Other; Categorical Analysis; GMR = 0.31, 90% CI 2-sided [0.25 to 0.39] — GMR = GM for Moderate RI / GM for Healthy Controls
Statistical Analysis 2: Comparison: [Part 1] Severe RI; Test type: Other; Categorical Analysis; GMR = 0.10, 90% CI 2-sided [0.07 to 0.16] — GMR = GM for Severe RI / GM for Healthy Controls

23. Primary Outcome: [Parts 1 and 2] Estimated CLr of Gefapixant 50 mg in Participants With BSA-Normalized eGFR (Regression Analysis)
Description: CLr values of plasma gefapixant based on BSA-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of CLr were natural log-transformed and evaluated with a linear fixed-effects model containing BSA-normalized eGFR as a continuous variable. The back transformed mean CLr and corresponding 95% CI were predicted at the midpoint of the BSA-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Parts 1 and 2 - Predose and at 0-12 hrs, 12-24 hrs, and 24-48 hrs post dose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. This population was used for regression analysis of the BSA-normalized CLr of gefapixant 50 mg. Renal clearance could not be assessed for participants with ESRD.
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6
L/hr | 1.49 [1.13 to 1.97] | 0.997 [0.711 to 1.40] | 5.95 [3.97 to 8.91]

24. Primary Outcome: [Parts 1 and 2] Estimated CLr of Gefapixant 50 mg in Participants With BSA Non-Normalized eGFR (Regression Analysis)
Description: CLr values of plasma gefapixant based on BSA non-normalized eGFR for participants with moderate RI, severe RI, or normal renal function (i. e., Healthy Controls) were estimated using regression analysis. Individual values of CLr were natural log-transformed and evaluated with a linear fixed-effects model containing BSA non-normalized eGFR as a continuous variable. The back transformed mean AUC0-inf and corresponding 95% CI were predicted at the midpoint of the BSA non-normalized eGFR range for each group (45 mL/min, 22.5 mL/min, and 139 mL/min for moderate RI, severe RI, and healthy controls, respectively). Although no participants with mild RI were included in this study, their BSA non-normalized eGFR estimates were predicted at midpoint 75 mL/min.
Time Frame: Parts 1 and 2 - Predose and at 0-12 hrs, 12-24 hrs, and 24-48 hrs post dose
Population: All participants in Parts 1 and 2 who were compliant with the study procedure and had available data were included. Renal clearance could not be assessed for ESRD participants. Participants originally assigned to the severe RI group were reassigned: 1 to the mild RI group (excluded from analysis), and 1 to the moderate RI group.
Measure: Mean (95% Confidence Interval); unit: L/hr
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 1] Healthy Controls
Number analyzed (Participants) | 7 | 4 | 6
L/hr | 1.36 [1.01 to 1.85] | 0.975 [0.677 to 1.41] | 5.53 [3.66 to 8.35]

25. Secondary Outcome: [Parts 1 and 2] Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants who experienced at least one adverse event (AE) was assessed. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure.
Time Frame: Parts 1 and 2 - Up to 29 days.
Population: All participants in Parts 1 and 2 who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2] ESRD | [Part 1 and Part 2] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 2 | 0 | 1

26. Secondary Outcome: [Parts 1 and 2] Number of Participants Discontinuing Study Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE was assessed. An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure.
Time Frame: Part 1 and 2 - Up to 15 days
Population: All participants in Parts 1 and 2 who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | [Part 1] Moderate RI | [Part 1] Severe RI | [Part 2] ESRD | [Part 1 and Part 2] Healthy Controls
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 29 days
Groups:
- MK-7264 50 mg: Moderate RI: Participants with moderate RI received a single oral dose of gefapixant 50 mg
- MK-7264 50 mg: Severe RI: Participants with severe RI received a single oral dose of gefapixant 50 mg
- MK-7264 50 mg: ESRD: Participants with ESRD requiring HD received a single oral dose of gefapixant 50 mg immediately after HD in Period 1, followed by a single oral dose of gefapixant 50 mg two hours prior to HD in Period 2. Between the Periods 1 and 2 MK-7264 dose administrations there was approximately a 7-day washout period with 3 dialysis sessions.
- Healthy Controls: Healthy control participants received a single oral dose of gefapixant 50 mg
Arm/Group | MK-7264 50 mg: Moderate RI | MK-7264 50 mg: Severe RI | MK-7264 50 mg: ESRD | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7264 50 mg: Moderate RI (N=6) | MK-7264 50 mg: Severe RI (N=6) | MK-7264 50 mg: ESRD (N=6) | Healthy Controls (N=6)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03108924/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03108924/SAP_001.pdf